CLINICAL TRIAL: NCT00969267
Title: The Effect of Auricular Point Stimulation on Obese Women: a Randomized Controlled Trial
Brief Title: The Effect of Auricular Point Stimulation on Obese Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Chung-Hua Hsu, vice superintendent, Taipei City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 98001-62-020
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Obesity
Keywords: ear acupuncture; obese; obese women; women
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Stimulation A (Experimental): with needle A stimulation
  Interventions: Other: ear-acupuncture A
- Stimulation B (Active Comparator): with stimulation
  Interventions: Other: stimulation B
- Stimulation C (Sham Comparator): without needle
  Interventions: Other: stimulation C

INTERVENTIONS:
Other: ear-acupuncture A — with needle stimulation
  Other Names: ear acupuncture needle
  Arms: Stimulation A
Other: stimulation B — with bread stimulation on ear acupuncture point
  Other Names: ear acupuncture bread
  Arms: Stimulation B
Other: stimulation C — without needle stimulation
  Other Names: placebo needle
  Arms: Stimulation C

SUMMARY:
The aim of the study is to examine whether the ear acupoint stimulation is effective on obese women.

DETAILED DESCRIPTION:
% change body weight, BMI, lipid profile, glucose and obese hormone.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-65 years women
* BMI>27 kg/mm
* Signed informed consent

Exclusion Criteria:

* Endocrine disease, e.g. thyroid disorder, pituitary disorder, and sex gland disorder.
* Heart disease, e.g. arrhythmia, heart failure, myocardial infarction, and patient with pacemaker.
* Allergy and Immunology disease.
* High aminotransferases ( Alanine, Aspartate > 80 IU/L) or high serum creatinine (> 2.5 mg/dL)
* Pregnant or lactating women.
* Childbirth within 6 months.
* Stroke or otherwise unable to exercise
* Management for weight control within 3 months.
* Any other conditions deemed unsuitable for trial as evaluated by the physician-in-charge.
* Endocrine disease

Ages: 16 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
% reducting of body mass index (BMI) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Hua Hsu, MD, PhD, Principal Investigator — Insitute of Traditional Medicine, National Yang Ming University
Locations (1):
- Branch of Chinese Medicine, Taipei City Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Hsu CH, Wang CJ, Hwang KC, Lee TY, Chou P, Chang HH. The effect of auricular acupuncture in obese women: a randomized controlled trial. J Womens Health (Larchmt). 2009 Jun;18(6):813-8. doi: 10.1089/jwh.2008.1005. PMID 19445642
- [Background] Hsu CH, Hwang KC, Chao CL, Lin JG, Kao ST, Chou P. Effects of electroacupuncture in reducing weight and waist circumference in obese women: a randomized crossover trial. Int J Obes (Lond). 2005 Nov;29(11):1379-84. doi: 10.1038/sj.ijo.0802997. PMID 15953937
- [Background] Hsu CH, Tsai TH, Kao YH, Hwang KC, Tseng TY, Chou P. Effect of green tea extract on obese women: a randomized, double-blind, placebo-controlled clinical trial. Clin Nutr. 2008 Jun;27(3):363-70. doi: 10.1016/j.clnu.2008.03.007. Epub 2008 May 12. PMID 18468736